CLINICAL TRIAL: NCT05950789
Title: Effect of Virtual Reality Application on Pain, Anxiety, and Vital Findings Due to Port Catheter Needle Insert Randomized Controlled Study
Brief Title: Port Catheter Needle Insert: A Virtual Reality Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Derya ÇINAR, Associate Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bakircay
Record Dates: First submitted 2023-06-12; First posted 2023-07-18 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Catheter Complications
Keywords: cancer; virtual reality; pain; anxiety; vital signs; Catheter Complications
MeSH Terms: conditions — Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality application group (Experimental): During the preparation stage of the port catheter injection attempt, the intervention group was given a calming video and music concert using virtual reality glasses.
  Interventions: Other: Virtual reality application
- Control (No Intervention): In the control group, no intervention was made other than the routine application.

INTERVENTIONS:
Other: Virtual reality application — During the preparation stage of the port catheter injection attempt, the intervention group was given a calming video and music concert using virtual reality glasses.
  With virtual reality glasses, patients watch three-dimensional video nature images, which we determined according to the patient's preference, accompanied by music. They put on the virtual reality glasses before the process started and removed them after the process was over.
  Arms: Virtual reality application group

SUMMARY:
The study was randomized controlled to examine the effect of virtual reality (VR) application on pain, anxiety, and vital signs associated with port catheter needle insertion. This study was conducted as a parallel-group, randomized controlled intervention study. The study was conducted with 84 cancer patients who came to Bursa Uludağ University outpatient chemotherapy unit for treatment between December 2022 and May 2023 and met the inclusion criteria. Patients undergoing port catheterization were randomly assigned to the intervention (n=42) and control (n=42) groups. During the preparation stage of the port catheter injection attempt, the intervention group was given a calming video and music concert using virtual reality glasses. In the control group, no intervention was made except the routine application.

DETAILED DESCRIPTION:
The purpose and rationale of the study were explained to the patients who met the inclusion criteria. Written informed consent was obtained from the patients who agreed to participate in the study. Patients were assigned to the intervention and control groups by simple randomization. The data of the study were collected simultaneously from both groups.

Standard care was applied to both groups during the port needle intervention procedure. Patients assigned to the intervention group were given standard care and VR application. The State Anxiety Scale was administered to the patients in both groups before the port catheter insertion procedure. Blood pressure, heart rate, respiratory rate, and oxygen saturation were measured and vital signs were recorded in the follow-up chart. The patients in the intervention group were informed by the researcher about the use of VR glasses and viewing the images. The contents of the VR images were shown to the patients on the smartphone and one of the images was presented to their preferences. Afterward, the patient was seated in the chair where he would receive chemotherapy, and VR glasses and headgear were put on. From the moment the position was given, the images preferred by the patients were applied to the VR application, which lasted for an average of 3 minutes, through VR glasses throughout the procedure. After the procedure was completed, the VR glasses were removed. Then, the State Anxiety Inventory, one of the data collection tools, was administered to the patients again. Visual Analogue Scale was used to determine the pain level of the patients due to the needle insertion procedure for the port catheter. After the procedure was completed, the patient's blood pressure, heart rate, respiratory rate, and oxygen saturation were measured again, and vital signs were recorded in the follow-up chart.

ELIGIBILITY:
Inclusion Criteria:

* Receiving active chemotherapy
* Those with a diagnosis of stage I-II and III cancer
* Those who volunteered to participate in the research
* With the implantable venous port catheter
* Those who will use virtual reality glasses for the first time

Exclusion Criteria:

* With metastases
* Receiving anxiolytic drug therapy
* Receiving antidepressant medication
* Communication, hearing, and vision problems
* Having any psychiatric disorder
* Using any analgesic drug at least 8 hours before
* Those with migraine, vertigo, active nausea-vomiting, headache, dizziness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
The State Anxiety Inventory | up to 24 hours
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Öner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
Vital signs chart-I | up to 24 hours
  It is applied to record patients by measuring systolic pressure (mmHg) at pre-intervention and post-intervention.
Vital signs chart-II | up to 24 hours
  It is applied to record patients by measuring diastolic pressure (mmHg) at pre-intervention and post-intervention.
Vital signs chart-III | up to 24 hours
  It is applied to record patients by measuring heart rate/ minute at pre-intervention and post-intervention.
Vital signs chart-IV | up to 24 hours
  It is applied to record patients by measuring respiratory rate/ minute at pre-intervention and post-intervention.
Vital signs chart-V | up to 24 hours
  It is applied to record patients by measuring oxygen saturation (%) at pre-intervention and post-intervention.
Visual Analog Scale | up to 24 hours
  VAS is a scale developed by Price et al. and measures the severity of pain in the patient. VAS is a 10 cm long vertical or horizontal scale with two different names (0=no pain, 10=most severe pain). An increase in the score obtained from the scale in the evaluation indicates an increase in pain.
  It is applied to determine the severity of pain in patients at immediately after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Derya ÇINAR, Assoc. prof., Principal Investigator — İzmir Bakircay University
Locations (1):
- İzmir Bakırçay University, Izmir, Turkey (Türkiye)